CLINICAL TRIAL: NCT04414215
Title: Cognitive Training for Emotion Regulation in Psychotic Disorders
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Georgia (Other)
Responsible Party: Principal Investigator, Gregory Paul Strauss, Associate Professor, University of Georgia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 00001377
Record Dates: First submitted 2020-05-26; First posted 2020-06-04 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Schizophrenia; Schizo Affective Disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Intervention Model Description: A double blind design will be used, where participants will be randomly assigned to placebo or emotional working memory training
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive training (Experimental): Emotional working memory training
  Interventions: Behavioral: Emotional working memory training
- Placebo training (Placebo Comparator): Placebo working memory training
  Interventions: Behavioral: Placebo working memory training

INTERVENTIONS:
Behavioral: Emotional working memory training — Participants will complete an emotional working memory n-back training program that progressively increases difficulty and has been shown to enhance prefrontal activity in a non-psychiatric sample
  Arms: Cognitive training
Behavioral: Placebo working memory training — Working memory training that does not involve emotional stimuli using an N-back training program
  Arms: Placebo training

SUMMARY:
The current study examines the efficacy of a cognitive training intervention for improving emotion regulation in psychotic disorders. it is hypothesized that the cognitive training program will enhance prefrontal activation, leading to enhanced emotion regulation.

DETAILED DESCRIPTION:
Psychotic disorders are serious and debilitating mental illnesses that incur substantial suffering for patients and present major challenges to our health care system. Difficulties with emotion regulation (i.e., the ability to control the emotion response using strategies) significantly predict the development and maintenance of psychotic symptoms and poor community-based functional outcomes. Recent neuroimaging research indicates that hypofrontality may underlie these deficits. Unfortunately, there is no accepted technique for remediating these emotion regulation abnormalities in psychotic disorders. Recent advances from the field of cognitive neuroscience provide hope for a resolution to this critical unmet need in psychotic disorder therapeutics, demonstrating that brief computerized cognitive training interventions are capable of improving emotion regulation ability by targeting neural activation in the prefrontal cortex. The goal of the proposed project is to determine whether an emotional working memory cognitive training program is effective for remediating emotion regulation abnormalities and associated clinical outcomes in people with psychotic disorders. Outpatients with psychotic disorders will be randomly assigned to either an emotional working memory training (n = 35) or placebo (P: n = 35) cognitive training control intervention delivered via an app on a smart phone for 30 days. The primary aim is to determine whether the emotional working memory intervention successfully engages the target mechanism and enhances prefrontal activation on a non-trained emotion regulation transfer task beyond a pre-specified effect size criterion. Results will also be used to determine the treatment duration (15 vs. 30 days) that most effectively and efficiently improves the target.

ELIGIBILITY:
Inclusion Criteria:

* diagnostic and statistical manual fifth edition diagnosis of schizophrenia or schizoaffective disorder
* 18-60 years old
* speaks English
* premorbid intelligence quotient > 70
* clinically stable as indicated by no antipsychotic medication changes in the last month or if on depot, no change in the past 2 months.

Exclusion Criteria:

* history of intellectual disability or neurological disorder
* history of traumatic brain injury with loss of consciousness > 10 minutes or behavioral sequelae
* substance use disorder within the last 6 months (other than nicotine)
* 4) endorsement of MRI exclusion factors

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Prefrontal blood oxygen level dependent activation in the prefrontal cortex | Change from baseline to 15 days or 30 days
  blood oxygen level dependent change in the prefrontal cortex as measured using functional magnetic resonance imaging. This will be calculated as a change from baseline to follow-up on the contrast score (unpleasant passive viewing condition - reappraisal) on the emotion regulation reappraisal task

CONTACTS AND LOCATIONS:
Locations (1):
- University of Georgia, Athens, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be uploaded to the National Institute of Mental Health Data Archive
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 1 year after study completion for 1 year
Access Criteria: The National Institute of Mental Health Data Archive request